CLINICAL TRIAL: NCT00168051
Title: A Single Dose, Randomized, 2-Period Crossover Study in Patients With Hemophilia A to Evaluate the Pharmacokinetics of ReFacto (B-domain Deleted Recombinant Human Factor VIII (BDDrFVIII) and Advante (a Full-length Recombinant Factor VIII (FLrFVIII)
Brief Title: Study Comparing Blood Levels of ReFacto and Advante in Hemophilia A
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3082A-101711
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2013-02

CONDITIONS: Hemophilia A
Keywords: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII SQ

INTERVENTIONS:
Drug: ReFacto
Drug: Advante

SUMMARY:
The purpose of the study is to compare the pharmacokinetic parameters of ReFacto and Advate, using the chromogenetic substrate assay to measure plasma Factor VIII activity in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A
* Previously treated patients with at least 150 exposure days to any Factor VIII product

Exclusion Criteria:

* Hypersensitivity to any recombinant Factor VIII product
* History of or current Factor VIII inhibitor
* Bleeding episode or other reason requiring Factor VIII treatment within 3 days of study

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measurement of area under the plasma Factor VIII activity in plasma versus time curve for 48 hours.

SECONDARY OUTCOMES:
Number of subjects who experience any adverse event or develop Factor VIII inhibitor at study termination, 48 hours post dosing and/or at the final study visit within seven days of the 2nd period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, MedInfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For New Zealand, medinfo@wyeth.com; Trial Manager, Principal Investigator — For UK, ukmedinfo@wyeth.com
Locations (13):
- United States (4):
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Iowa City, Iowa
  - New Orleans, Louisiana
- Brussels, Belgium
- Paris, France
- Germany (2):
  - Berlin
  - Münster
- Milan, Italy
- Netherlands (2):
  - Amsterdam
  - Utrecht
- Christchurch, New Zealand
- Manchester, United Kingdom